CLINICAL TRIAL: NCT00309192
Title: Efficacy and Safety of Intravitreal Triamcinolone as Treatment of the Diffuse Diabetic Macular Edema
Brief Title: Efficacy and Safety Study of Intravitreal Triamcinolone to Treat Diffuse Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-001385-14; PI071701
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2009-01

CONDITIONS: Diabetes Mellitus; Macular Edema
Keywords: Diabetes, Macular Edema, Triamcinolone
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Triamcinolone Acetonide; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Triamcinolone acetonide + Grid Laser
  Interventions: Drug: Triamcinolone Acetonide; Procedure: Grid laser
- 2 (Sham Comparator): Sham procedure + Grid laser
  Interventions: Procedure: Grid laser; Procedure: Sham Injection

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Intravitreal Injection 4mg single dose
  Other Names: Trigon Depot
  Arms: 1
Procedure: Grid laser — Grid laser as specified in ETDRS
Procedure: Sham Injection — Simulation procedure for triamcinolone injection
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether intravitreal injection of Triamcinolone Acetonide is effective in the treatment of Clinically Significant Diffuse Macular Edema due to Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus and its complications represent nowadays an important issue in Public Health terms. The WHO expectations indicate that around 2025 the European population with diabetes will reach about 12%, and it has been estimated that the percent in the USA will be around 10% (King, 1995).

The severe complications of proliferant diabetic retinopathy and its disastrous effects on vision seem to be solved with retinal panphotocoagulation. The most relevant issue regarding diabetes´ ocular complications seems to be macular edema. We define macular edema as retinal thickening between 1500 microns central to fovea. It is found in about 10% diabetics, of whom about 40% will have an important visual acuity loss (Klein, 1984) In our environment, diabetes retinopathy affects nearly 21% of all the diabetics, and among them, about 6% has a clinically significant macular edema (Lopez, 2001).

Until now the only treatment available with proved efficacy for diffuse edema was grid photocoagulation, stablished as standard treatment since the publication of results from "Early Treatment Diabetic Retinopathy Study" (Olk 1990). A maximum 3 laser treatments with 3 to 4 months intervals between treatment has been accepted.

Nevertheless, the results with the treatment haven´t been considered satisfactory as the main aim is to preserve visual function, and only 15% of the patients get any improvement (Mc Donald, 1985).

Because of that more alternatives have been studied, among them victrectomy and intraocular corticosteroyd injections. Though, vitrectomy seems to provide significative improvements only if the patient has a thickened posterior hyaloid able to make a traction over the macular area (Tachi, 1996) and that doesn´t happen in the majority of diabetic patients.

The identification of Vascular Endothelial Growth Factor (VEGF) as the main responsible agent of angiogenesis and its role in the pathogenia of diabetic macular edema has opened new approach methods in the treatment of this complication (Adamis 1994). This factor, also known as Vascular Permeability Factor (VPF), interacts with "tight junctions" of retinal endothelial cells, producing a disruption of hematoretinal barrier.

It is known that corticosteroids are not only the more powerful antiangiogenetic agents, but are also capable of reversing the effects mentioned before over the retinal endothelial by acting at phosphorilation and expression of tight-junctions´ proteins. They also inhibit VEGF expression (Fisher 2001).

It seems logical that its use has been proposed in the treatment of this diabetes complication. Though, its side effects, either local or systemical, and its intraocular biodisponibility issues have obligated the use of intravitreal administration.

In 2001 was published the first work about intravitreal triamcinolone after vitrectomy in proliferative diabetes retinopathy patients, in an attempt to reduce the inflammatory response what sometimes occurs in these patients after surgery (Jonas, 2001). A series of 29 eyes shows a good tolerance of the drug administered this way.

The next year, and after the presentation at ARVO meeting, some other authors present a prospective work without control group with 16 eyes of patients who have been injected triamcinolone acetonide after grid laser failure, applied according to ETDRS criteria. The results show a visual acuity improvemente and a reduction of macular edema evaluated with ocular coherence tomography, with an effect loss in a 6 months interval (Martidis, 2002).

Since then more clinical series have been published, but yet without any prospective, randomized and control group studies done.

These series seem to show a positive effect of triamcionlone either in 25 mg dosage (Jonas, 2002) or 4 mg dosage.

It is remarkable that the majority of the studies have been published by Heidelberg Group, although series from other authors are also being published (Massin, 2004).

There has also been published side effects as ocular hypertension and endophthalmitis, that seem not to be infectious in the majority of the cases (Roth, 2003) but due to its high prevalence they need to be studied in depth.

This approach is being taken by some pharma industries with variations; intraocular controlled liberation implants of fluocionola acetonide or dexametasone biodegradable implants have been developed (Jaffe 2000).

It is also being investigated the potential effect of Anecortave acetate, a cortisol derivate, and there are also some other alternatives under research: VEGF inhibitors as adaptamers, andibodies or fragments, PKC inhibitors or angiopoiteins, some of which are currently being evaluated in Phase III Clinical Trials.

Despite the lack of clinical trials similar to the one proposed here, the topic has provoked a lot of interest in the international and national ophthalmological community and there are evidences of some of these treatments being used in our country.

Comparisons:

Study Group: TRIGON DEPOT (Bristol Mayers Squibb Labs) 4 mg intravitreal injection followed by ETDRS grid laser technique.

Control Group: ETDRS grid laser technique.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes.
* Mild-moderate diabetes retinopathy.
* Diffuse clinically significant macular edema (demonstrated by angiofluoresceingraphy, associated or not to cystic changes).
* Age between 50 to 75 years.
* Foveal thickening greater than 300 microns tested with Optical Coherence Tomography (OCT).
* Visual acuity better than 0,05.
* None of the exclusion criteria.
* Informed consent signed.
* Data protection consent signed.

Exclusion Criteria:

* Bad metabolic control in recruitment stage (as criteria from Endocrinology Department of each Center) or Glicosilated Hemoglobine greater than 9%.
* Uncontrolled hypertension. Greater than 150/90.
* Systemic treatment with oral corticosteroids, diuretics or immunosupressors 3 months before or during the study.
* Record of ocular hypertension induced by corticosteroids.
* Glaucoma or ocular hypertension.
* Unbalanced heart failure.
* Any other pathology that could cause macular edema.
* Associated ischemic maculopathy. (Parafoveal avascular area thickening greater than 1000 microns)
* Patients with Clinically Significant Macular Edema with posterior hyaloid thickening or macular traction in biomicroscopy or OCT.
* Patients with panretinophotocoagulation.
* Patients that will probably need a panretinophotocoagulation during the study (6 to 12 months).
* Record of ocular herpes infection.
* Lens opacification that may interfere with clinical, photographical or OCT examinations.
* Toxoplasmosis, active or not in the study eye.
* Vitrectomy in either eye.
* Record of Central Serose Coroidopathy.
* Pseudophakic patients with less than 6 months since surgery.
* Patients with any other situation that may interfere in study completion based in Investigator´s opinion.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Visual acuity stabilization or improvement 6 months after treatment. | 6 months
Macular edema reduction or stabilization 6 months after treatment. | 6 months

SECONDARY OUTCOMES:
Safety of the treatment. | 6 months
Tolerance of the treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Pastor Jimeno, MD, PhD, Study Director — IOBA - Instituto de Oftalmobiología Aplicada - Universidad de Valladolid
Locations (7):
- Spain (7):
  - INGO - Instituto Galego de Oftalmoloxia, Santiago de Compostela, La Coruña
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Instituto Oftalmológico de Alicante, Alicante
  - Hospital de la Vall D´Hebrón, Barcelona
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital General Universitario Reina Sofía, Murcia
  - IOBA - Instituto Universitario de Oftalmobiología Aplicada, Valladolid